CLINICAL TRIAL: NCT00348491
Title: A Randomized, Double-blind, Double-dummy, Parallel Group, Single-center Study Evaluating the Analgesic Effect of Single Doses of Lumiracoxib 400 mg, Celecoxib 400 mg and Placebo in the Treatment of Post-dental Surgery Pain
Brief Title: Efficacy of Lumiracoxib in Relieving Moderate to Severe Post-dental Surgery Pain, Compared to Both Placebo and Celecoxib
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2474
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pain
Keywords: Dental surgery; acute pain; lumiracoxib; celecoxib; Moderate to severe pain following dental surgery
MeSH Terms: conditions — Pain; Acute Pain | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study will assess the safety and efficacy of lumiracoxib 400 mg in relieving moderate to severe post-dental surgery pain, compared to both placebo and celecoxib 400 mg.

ELIGIBILITY:
Inclusion Criteria:

* Requiring extraction of two or more partially impacted or fully bony impacted third molars. At least one of the extractions must be mandibular
* Moderate to severe post-dental surgery pain intensity (as rated by the patient on the categorical pain intensity scale within five hours of surgery

Exclusion Criteria:

* Evidence or history of any cardiac and cerebral thrombotic/ ischemic diseases and/ or events

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 364
Dates: Start 2006-02; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Superiority of a single dose of lumiracoxib 400 mg compared to placebo and celecoxib 400 mg based on a Summed (time weighted) Pain Intensity Difference calculated over 0-8 hours post-dose (SPID-8)

SECONDARY OUTCOMES:
Evaluate efficacy of a single dose of lumiracoxib 400 mg compared to placebo and to celecoxib 400 mg in relieving post dental surgery pain with respect to the following secondary efficacy variables:
Time-specific Pain intensity Difference (PID) based on the categorical scale, Pain Relief (PR) based on the categorical scale, and Pain Relief Intensity Difference (PRID) (sum of PID and PR based on categorical scales) at time-points up to 24 hours after
Time-specific PID based on VAS at time-points up to 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (1):
- Dental Research Clinic, Austin, Texas, United States

REFERENCES:
- [Result] Fricke J, Davis N, Yu V, Krammer G. Lumiracoxib 400 mg compared with celecoxib 400 mg and placebo for treating pain following dental surgery: a randomized, controlled trial. J Pain. 2008 Jan;9(1):20-7. doi: 10.1016/j.jpain.2007.08.004. Epub 2007 Oct 15. PMID 17933588